CLINICAL TRIAL: NCT07400354
Title: A Study on the Assessment of the Efficacy of PD-1 Monoclonal Antibody Combined With Chemotherapy in Metastatic Gastric Cancer Based on Gut Microbiota
Brief Title: The Efficacy of PD-1 Monoclonal Antibody Combined With Chemotherapy in Metastatic Gastric Cancer Based on Gut Microbiota
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhu, chief physician, Fudan University
Other Study IDs: MGC-FLORA
Record Dates: First submitted 2026-01-25; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Gastric Cancer; Gut Microbiota
MeSH Terms: conditions — Stomach Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study, no intervention — Observational study, no intervention

SUMMARY:
This study is designed as a single-center, open-label, phase II exploratory trial. Patients with advanced or locally advanced gastric cancer who have not received chemotherapy or immunotherapy before are eligible for inclusion. They will receive a first-line two-drug combination chemotherapy regimen (FOLFOX, XELOX, or SOX, determined by the attending physician) in combination with a PD-1 monoclonal antibody (nivolumab, sintilimab, tislelizumab, or pembrolizumab, determined by the attending physician). Fruquintinib can be added on this basis (only for patients enrolled in the HMPL-013-SH-GC103 study). The aim is to evaluate whether the gut microbiota has a predictive role in the efficacy of immunotherapy combined with chemotherapy for metastatic gastric cancer. A total of 100 patients will be enrolled in the study.

Gut microbiota will be measured at the following three time points:

1. Within 3 days before the first chemotherapy (designated as time 0)
2. Within 3 days before the third chemotherapy (designated as time 1)
3. After the sixth chemotherapy cycle, or within 1 week after disease progression if it occurs within the sixth cycle (designated as time 2)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, gender not restricted;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score 0-2, with -an expected survival period of more than 3 months;
* Metastatic or locally advanced gastric cancer confirmed by cytology or histopathology;
* Laboratory test data within 7 days before screening (including 7 days) should meet the following requirements: neutrophil count ≥ 1.5×109/L, platelet count ≥ 80×109/L, hemoglobin ≥ 80g/L, total serum bilirubin ≤ 1.5 times the upper limit of normal (ULN); ALT and AST ≤ 2.5 x ULN, if liver metastasis is present, ALT and AST ≤ 5 x ULN; albumin ≥ 30g/L; serum creatinine ≤ 1.5 x ULN or creatinine clearance rate (CCr) ≥ 60ml/min.
* At least one evaluable lesion (according to RECIST 1.1 criteria);
* No previous palliative chemotherapy and planned for first-line immunotherapy (nivolumab, sintilimab, tislelizumab, pembrolizumab as recommended by guidelines, specifically determined by the attending physician) combined with chemotherapy (FOLFOX, XELOX, SOX, specifically determined by the attending physician), and combination with fruquintinib is allowed (only for patients enrolled in the trial with the number HMPL-013-SH-GC103);
* The subject (or their legal representative/guardian) must sign the informed consent form, indicating that they understand the purpose of this study, are aware of the necessary procedures, and are willing to participate in this study.

Exclusion Criteria:

* Pregnant or lactating women, and women of childbearing age who have not taken adequate contraceptive measures;
* Patients with a history of other malignant tumors within 5 years, except for those with a history of cured cervical carcinoma in situ or non-melanoma skin cancer; Patients with primary brain tumors or central nervous system metastases that are not under control, and those with obvious intracranial hypertension or neuropsychiatric symptoms;
* Patients with the following severe or uncontrolled diseases: severe heart disease, unstable condition despite treatment, myocardial infarction, congestive heart failure, unstable angina pectoris, significant pericardial effusion or unstable arrhythmia within 6 months before enrollment; definite neurological or psychiatric disorders, including dementia or epileptic seizures; severe or uncontrolled infections; active disseminated intravascular coagulation, or patients with obvious bleeding tendencies;
* Patients with significant damage to important organs;
* Patients with pleural effusion or ascites causing respiratory syndrome (≥CTCAE grade 2 dyspnea) requiring local treatment;
* Other conditions where the investigator deems the patient unsuitable for participation in this trial;
* Patients who have been taking probiotics or antibiotics for a long time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2027-03-14 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The gut microbiota predicts progression-free survival (PFS) | the duration from the date of randomization to any documented tumor progression or death due to any cause，assessed up to 36 months
  The gut microbiota predicts progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
We would like to share data if request.